


# Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the DVR® Plating System (Implant and Instrumentation)

A Retrospective Consecutive Series Study

Revision 1 08/05/2019 NCT04653051

#### STUDY SPONSOR

Zimmer GmbH
Sulzerallee 8
P.O. Box
CH-8404 Winterthur
Switzerland
Tel. +41 (0)58 854 80 00






Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and

Clinical Benefits Data of the DVR® Plating System (Implant and

Instrumentation) – A Retrospective Consecutive Series Study

**CIP ID:** MDRG2017-89MS-14T

Sponsor: Zimmer GmbH

Manufacturer: Biomet Trauma, Warsaw, Indiana, USA

**Objectives:** The objective of this retrospective PMCF study is to collect data confirming

safety, performance and clinical benefits of the DVR Plating System (implant

and instrumentation) when used for the treatment of wrist fractures.

The primary objective is the assessment of performance by analyzing fracture

healing.

The secondary objectives are the assessment of safety by recording and

analyzing the incidence and frequency of complications and adverse events.

Relation of the events to implant, instrumentation and/or procedure should be

specified. Patients' outcomes will also be assessed.

**Population:** Consecutive series of subjects implanted with one of the DVR Plating System

according to the approved/cleared indications. Inclusion/exclusion criteria are

in accordance to the indications and contraindications in the IFU. The devices

included in the study will be the ones used in accordance with their IFU and/or

Zimmer Biomet's approved labeling.

Inclusion/Exclusion Criteria

Inclusion Criteria:

All subjects must have been implanted with one of the DVR Plates

according to the approved indications.






| | Exclusion Criteria: |
|---|---|
| | - Off-label use |
| | - Cases where there is an active infection |
| | - Conditions which tend to retard healing such as, blood supply limitations, previous infections, etc |
| | - Insufficient quantity or quality of bone to permit stabilization of the fracture |
| | - Conditions that restrict the patient's ability or willingness to follow postoperative instructions during the healing process |
| | <ul> <li>Foreign body sensitivity – where material sensitivity is suspected,<br/>appropriate tests should be conducted and sensitivity ruled out prior<br/>to implantations</li> </ul> |
| | - Cases where the implant(s) would cross open epiphyseal plates in skeletally immature patients |
| | - Cases with malignant primary or metastatic tumors which preclude adequate bone support or screw fixations, unless supplemental fixation or stabilization methods are utilized |
| Study Design: | Single-center, Retrospective, Consecutive series |
| Clinical Phase: | Post-market |
| Number of<br>Subjects: | 115 cases (in 111 patients) implanted with the DVR Plating System: |
| Length of Study: | 12 months overall: |
| | - Ethics Committee approval, patients' identification, consent and enrollment into the study |
| | - Collection of baseline information available in medical notes from the pre-OP condition to the immediate post-OP and last consultation visit |
| | - Conduct follow-up phone calls, data collection, analysis, and final report |













# DVR Wrist Plates (and respective instrumentation) **Dorsal Plate Radial Styloid Plate Ulna Plate** DVR Volar Rim Plates (and respective instrumentation) **DVR Volar Rim DVR Volar Rim Narrow Score:** Patient-Rated Wrist Evaluation Score (PRWE) **Documentation:** Paper / electronic **Statistical Analysis:** Data collected in the study will be summarized descriptively. Continuous data (e.g. age) will be summarized through means, medians, standard

deviation, minimum, maximum and 95% confidence intervals (CIs).



#### Revision 1

## **Clinical Investigation Plan**


Categorical data (e.g. gender) will be summarized using counts, percentages and 95% confidence limits. Summaries of fracture healing and osteotomy rates, implant related revision rates and complication data will be presented as frequencies and percentages.

#### References

1. Clinical Investigation of medical devices for human subjects – Good Clinical practice. ISO 14155:2011.